CLINICAL TRIAL: NCT03595722
Title: High Intensity Focused Ultrasound as a Treatment for Rectal and Pelvic Cancers - Laboratory and Clinical Feasibility Studies
Brief Title: Exploring HIFU as a Treatment for Rectal and Other Pelvic Cancers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Collaborators: SonaCare Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18SM4430
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Rectal Cancer; Rectal Neoplasms; Pelvic Cancer; Endometrial Cancer; Cervical Cancer
Keywords: Pelvic cancer; rectal cancer; HIFU; QoL; complications
MeSH Terms: conditions — Rectal Neoplasms; Pelvic Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early rectal cancer (Experimental): Patients with early rectal cancer undergoing a treat and resect pathway - patients will be treated with high intensity focused ultrasound 7-10 days prior to the surgical resection of their rectal cancer
  Interventions: Device: High Intensity Focused Ultrasound
- Late pelvic cancer (Experimental): Patients with late pelvic (rectal, endometrial, cervical) cancer will undergo a treat and observe pathway - patients will be treated with high intensity focused ultrasound and their response will be observed
  Interventions: Device: High Intensity Focused Ultrasound

INTERVENTIONS:
Device: High Intensity Focused Ultrasound — High intensity focused ultrasound to rectal/pelvic cancer

SUMMARY:
The hypothesis of the study is that high intensity focused ultrasound (HIFU) can be used safely to treat rectal and pelvic cancer. The study consists of two trials exploring the use of HIFU in rectal and pelvic cancer to establish the safety and potential efficacy of HIFU in this instance.

The first trial is a feasibility study looking at patients with early rectal cancer. We aim to recruit thirty patients with early rectal cancer who are due to undergo an operation to remove their cancer. After recruiting and consenting them for the trial, we will treat their rectal cancer with HIFU. Approximately one week after treatment they will undergo their normal cancer operation. This will allow us to demonstrate the safety of HIFU as a treatment for rectal cancer and evaluate the changes in rectal and surrounding tissue under the microscope after the cancer is treated with HIFU. In addition, we will monitor patients for any complications and the impact this treatment has on their quality of life. We will monitor the response of various markers for cancer with blood tests.

The second trial aims to evaluate the treatment of a cohort of patients with inoperable rectal cancer. We aim to recruit thirty patients with either inoperable pelvic cancers - rectal, cervical or endometrial, or cancers that have returned after previous operations. We will offer these patients treatment of their cancer using HIFU. We will monitor the symptoms they experience and impact on their quality of life both before and at multiple time points after the treatment with HIFU. We will compare MRI scans before and after treatment to evaluate the effect HIFU has in reducing the size of the cancer. We hope to show that using HIFU in this group of patients can be both effective and lead to an improvement in both their symptoms and quality of life.

DETAILED DESCRIPTION:
The hypothesis of this study is that high intensity focused ultrasound (HIFU) can be safely and effectively used to treat rectal and advanced pelvic cancers. This study is composed of two feasibility trials to evaluate the safety and efficacy of use in HIFU in early rectal cancer and late pelvic cancer.

The first trial will involve a cohort of 30 patients with early rectal cancer. They will have full work up as per normal care including history, examination, bloods, endoscopy and imaging (CT and MRI scan). Once eligibility has been confirmed, patients will be approached and offered to be enrolled in the study. Once successfully recruited, they will be admitted transrectal HIFU using the Sonatherm (Sonacare Medical, Charlotte, North Carolina, USA) device under general anaesthetic with monitoring for toxicity. Baseline quality of life questionnaires will be filled in by patients prior to HIFU to establish their symptoms prior to treatment. Patients will be admitted for treatment and observed overnight. They will then complete the same questionnaires at two and seven days post HIFU. Blood tests will be taken one week after HIFU administration to monitor levels of tumour markers and inflammatory markers. One week after their HIFU treatment, the patients will undergo their total mesorectal excision (TME) to remove their cancer as per normal treatment protocol. The specimen will be examined to evaluate the histological changes in the tumour and surrounding tissues created by the HIFU. We will be able to quantify the effect of HIFU on the rectal cancer and evaluate for possible thermal damage to surrounding tissues.

Potential patients will be identified during multidisciplinary team (MDT) meetings which include surgeons, radiologists, oncologists and cancer nurse specialists. The team will confirm eligibility and suitability prior to patient recruitment to ensure there is no negative effect on overall patient care due to their involvement in the trial.

The Sonatherm™ systems used ultrasound visualisation to monitor and regulate the HIFU delivery. This allows tissue response to HIFU to be monitored via echogenic changes seen during coagulative necrosis. The strong correlation between echogenic changes and tissue destruction will allow us to alter the power settings if needed to achieve suitable ablation of the target area. A video record of the ultrasound and ablation will be reviewed by the team to evaluate the quality of the ablation performed.

The trial will run for approximately 1 month for each patient: from recruitment into the study to the resection of the cancer. The HIFU dose will cover the entire tumour, the rectal wall, and a 5 mm margin of tissue surrounding the tumour. It is anticipated that all tissue exposed to HIFU, including the rectal wall, will be part of the coagulative necrosis. Antibiotic prophylaxis will be given for five days to reduce the risk of abscess formation and sepsis. Patients will be followed up on day 2 post HIFU and the day of their TME to assess their response to treatment and any complications that develop. Post resection the patients will be followed up as per the normal local guidelines following surgical excision of rectal cancer. They will have their quality of life post resection assessed by completing questionnaires 30 days post resection.

The second part of the study will involve a cohort of 30 patients with either locally advanced pelvic cancer (rectal, endometrial or cervical) or locally recurrent disease. These patients will be unsuitable for operative intervention or any further chemo-radiotherapy treatment. They will have full work up as per normal care including history, examination, bloods, endoscopy and imaging (CT and MRI scan). Once eligibility has been confirmed, patients will be approached and offered to be enrolled in the study. Once successfully recruited, they will be admitted intracavity HIFU using the Sonatherm™ device under general anaesthetic with monitoring for toxicity. Baseline quality of life questionnaires will be filled in by patients prior to HIFU to establish their symptoms prior to treatment. Patients will be admitted for treatment with HIFU and observed overnight to monitor for any toxicity related to treatment with HIFU. Antibiotic prophylaxis will be given for five days to reduce the risk of abscess formation and sepsis. Patients will be followed up closely to monitor for toxicity and any changes in symptom control/quality of life. Patients will complete the same pre-operative questionnaires at multiple time-points post HIFU treatment. Questionnaires will be completed at seven, thirty, sixty and ninety days post HIFU, and three-monthly thereafter. This will enable us to accurately chart the change in quality of life and symptom control created by the HIFU treatment. Post-treatment imaging will be performed at between 3-4 weeks, as within this time frame the ablative effect (a necrotic area) as seen in prostate cancer treated by HIFU. This will allow comparison with pre-operative imaging to evaluate the effect of HIFU. A video record of the ultrasound and ablation will be reviewed by the team to evaluate the quality of the ablation performed.

Patients will be reviewed at regular intervals after treatment with HIFU to monitor the effect of HIFU on quality of life. Regular blood tests will be taken to monitor tumour markers and markers of systemic inflammation.

Potential patients will be identified during MDT meetings which include surgeons, radiologists, gynaecologists, oncologists and cancer nurse specialists. The team will confirm eligibility and suitability prior to patient recruitment. If felt appropriate by the MDT, patients may be offered a second application of HIFU as necessary.

The trial will run in two stages: the end of the first phase (for regulatory requirements) is defined as 30 days from the date that the last patient has completed trial therapy. The non-interventional follow-up stage will then commence in which patients are followed up for a minimum of 6 months or death.

ELIGIBILITY:
Inclusion Criteria:

Early rectal cancer arm:

1. Biopsy proven rectal cancer <15cm from anal verge
2. Targeted region ≤ 3cm in depth dimension, deepest region of tumour ≤ 3.5cm from organ/tissue surface accessible by the probe
3. Tumour accessible by the HIFU probe via suitable acoustic window
4. Early stage disease not requiring neo-adjuvant chemo radiotherapy prior to TME - T1/T2 but confirmed to require adjuvant chemotherapy
5. Ability to undergo an intraluminal ultrasound examination
6. World Health Organisation (WHO) Performance Status 0-3
7. Age ≥18 and fit for general anaesthetic and HIFU
8. For women of child bearing potential, not pregnant
9. No other serious uncontrolled concomitant illness likely to interfere with treatment or assessment
10. Written informed consent for treatment

Late pelvic cancer arm:

1. Biopsy proven rectal, vaginal, endometrial or cervical cancer (tumour <15cm from anal/vaginal verge)
2. Solid tumour/mass ≤ 3cm in depth dimension, deepest region of tumour ≤ 3.5cm from organ/tissue surface accessible by the probe
3. Lymph node(s) accessible by HIFU for which the primary clinical team advise intervention
4. Tumour accessible by the HIFU probe via suitable acoustic window
5. Partially fixed/unresectable disease and locally advanced disease (T3/T4)
6. Ability to undergo an intraluminal ultrasound examination
7. WHO Performance Status 0-3
8. Age ≥18 and fit for general anaesthetic and HIFU
9. For women of child bearing potential, not pregnant
10. No other serious uncontrolled concomitant illness likely to interfere with treatment or assessment
11. Written informed consent for treatment

Exclusion Criteria:

Early rectal cancer arm:

1. WHO performance status of 4
2. Uncontrolled cardiac, respiratory or other disease, or any serious medical or psychiatric disorder that would preclude anaesthetic or informed consent
3. Pelvic sepsis
4. Currently enrolled in any neo-adjuvant treatment trial that may induce tumour regression
5. Locally advanced disease - T3/T4 or patients who are not thought to require adjuvant therapy
6. Tumours above peritoneal reflection or below dentate line
7. Subjects with tumours lying < 1cm from sensitive structures/organs

Late pelvic cancer arm:

1. WHO performance status of 4
2. Uncontrolled cardiac, respiratory or other disease, or any serious medical or psychiatric disorder that would preclude anaesthetic or informed consent
3. Pelvic sepsis
4. Currently enrolled in any other palliative treatment trial that may confound results
5. Subjects with tumours lying < 1cm from sensitive structures/organs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2022-08-28 (Estimated); Study Completion 2022-08-28 (Estimated)

PRIMARY OUTCOMES:
Complications | 0-30 days
  Complications and toxicity of HIFU treatment

SECONDARY OUTCOMES:
Symptom control | 7-90 days
  Quality of life questionnaire responses
Histological tissue changes | 7-10 days
  Histological changes in tumour and surrounding tissue
Tumour marker changes | 7-90 days
  Changes in circulating tumour markers
Inflammatory marker changes | 7-90 days
  changes in circulating inflammatory markers
Radiological changes | 30 days
  MRI changes in tumour

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Murphy, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thuroff S, Chaussy C, Vallancien G, Wieland W, Kiel HJ, Le Duc A, Desgrandchamps F, De La Rosette JJ, Gelet A. High-intensity focused ultrasound and localized prostate cancer: efficacy results from the European multicentric study. J Endourol. 2003 Oct;17(8):673-7. doi: 10.1089/089277903322518699. PMID 14622488
- [Background] Hill CR, ter Haar GR. Review article: high intensity focused ultrasound--potential for cancer treatment. Br J Radiol. 1995 Dec;68(816):1296-1303. doi: 10.1259/0007-1285-68-816-1296. PMID 8777589
- [Background] Gelet A, Chapelon JY, Bouvier R, Souchon R, Pangaud C, Abdelrahim AF, Cathignol D, Dubernard JM. Treatment of prostate cancer with transrectal focused ultrasound: early clinical experience. Eur Urol. 1996;29(2):174-83. PMID 8647143
- [Background] Wu F, Wang ZB, Chen WZ, Bai J, Zhu H, Qiao TY. Preliminary experience using high intensity focused ultrasound for the treatment of patients with advanced stage renal malignancy. J Urol. 2003 Dec;170(6 Pt 1):2237-40. doi: 10.1097/01.ju.0000097123.34790.70. PMID 14634387
- [Background] Stewart EA, Gedroyc WM, Tempany CM, Quade BJ, Inbar Y, Ehrenstein T, Shushan A, Hindley JT, Goldin RD, David M, Sklair M, Rabinovici J. Focused ultrasound treatment of uterine fibroid tumors: safety and feasibility of a noninvasive thermoablative technique. Am J Obstet Gynecol. 2003 Jul;189(1):48-54. doi: 10.1067/mob.2003.345. PMID 12861137
- [Background] Monzon L, Wasan H, Leen E, Ahmed H, Dawson PM, Harvey C, Muhamed A, Hand J, Price P, Abel PD. Transrectal high-intensity focused ultrasonography is feasible as a new therapeutic option for advanced recurrent rectal cancer: report on the first case worldwide. Ann R Coll Surg Engl. 2011 Sep;93(6):e119-21. doi: 10.1308/147870811X592458. PMID 21929907